CLINICAL TRIAL: NCT00648310
Title: Is There A Synergic Effect Of Topical Oestrogens When Associated To Antimuscarinics In The Treatment Of Symptomatic Detrusor Overactivity
Brief Title: Topical Oestrogens and Antimuscarinics In The Treatment Of Detrusor Overactivity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Other Study IDs: local oestrogens 9/2003
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): arm 1: Tolterodine 4 mg once daily for 12 weeks
  Interventions: Drug: Tolterodine 4 mg
- 2 (Experimental): arm 2: Tolterodine 4 mg + local oestrogens once daily for 12 weeks
  Interventions: Drug: arm 2: Tolterodine 4 mg + local oestrogens once daily for 12 weeks

INTERVENTIONS:
Drug: Tolterodine 4 mg
  Arms: 1
Drug: arm 2: Tolterodine 4 mg + local oestrogens once daily for 12 weeks
  Arms: 2

SUMMARY:
Despite the great number of reports about the efficacy of oestrogens or antimuscarinics on OAB symptoms, so far no author has tried to investigate whether the concomitant administration of these two drugs, acting on two different pathophysiological mechanisms, could have a synergic effect reducing the rate of non-responders to treatment.

ELIGIBILITY:
Inclusion Criteria:

* All post-menopausal women with symptoms of overactive bladder and urodynamically proven pure detrusor overactivity

Exclusion Criteria:

* concomitant urodynamic stress incontinence
* documented recurrent urinary tract infections
* previous antimuscarinic treatment
* previous pelvic surgery
* concomitant systemic HRT
* history of breast or endometrial cancer
* neurological disease
* clinical contraindications to treatment with oestrogen or antimuscarinics
* patients included in other ongoing clinical trials

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-01; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology and Obstetrics - Università dell'Insubria, Varese, Italy

REFERENCES:
- [Derived] Serati M, Salvatore S, Uccella S, Cardozo L, Bolis P. Is there a synergistic effect of topical oestrogens when administered with antimuscarinics in the treatment of symptomatic detrusor overactivity? Eur Urol. 2009 Mar;55(3):713-9. doi: 10.1016/j.eururo.2008.06.051. Epub 2008 Jun 20. PMID 18584946